CLINICAL TRIAL: NCT03827122
Title: Botulinum Toxin A Injectable Solution in the Management of Bruxism
Brief Title: Botulinum Toxin A Injectable Solution in the Management of Bruxism: A Clinical Trial Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Baraa Abdulrahman, Master Resident in Oral Diagnostics, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC/IRB/2018/1247
Record Dates: First submitted 2019-01-11; First posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Nocturnal Bruxism
Keywords: Bruxism
MeSH Terms: conditions — Sleep Bruxism; Bruxism | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Single group with bruxism they will be injected in masster muscles bilaterally
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Group one (Experimental): Botx will be injection in masster muscles 20unit Botx (onabotulinumtoxinA) and visual pain scale will be taken before and after in four intervals 2,8,16,48 weeks
  Interventions: Drug: onabotulinumtoxinA

INTERVENTIONS:
Drug: onabotulinumtoxinA — Experimental group we will use BTX-A administration group. All patients (Male/Female) with bruxism associated with chronic pain in masseter muscles bilaterally Patients will have treatment with 20 units of BOTOX, (Allergan Inc.) per side will be injected at three points into masseter muscle bilaterally.
  Other Names: Botox Allergan

SUMMARY:
A Clinical Trial Study to investigate the potential performance of BTXA on masseter muscle on patient with nocturnal bruxism and to check the pain scale and share this clinical experience.

DETAILED DESCRIPTION:
Experimental group we will use BTX-A administration group. All patients (Male/Female) with bruxism associated with chronic pain in masseter muscles bilaterally participated in this study. The patients age 18-60 years. According to the diagnostic grading system of bruxism all subjects will have an assessment including a bruxism questionnaire (i.e., oral history taking with specific focus on bruxism habits) plus a clinical examination to evaluate bruxism signs and symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate to severe pain in relation to the masseter muscles and TMJ area related to bruxism during clinical examination.
2. Aged 20-60 patients.
3. Tooth-grinding sounds corroborated by family members or caregivers.
4. Cases where bruxism resulted in occlusal surface attrition of posterior teeth

Exclusion Criteria:

1. pain in the orofacial region,
2. insomnia,
3. known botulinum toxin allergy,
4. pregnancy,
5. neuromuscular disease,
6. bleeding disorders,
7. antibiotic therapy,
8. pulmonary disease that produced coughing during sleep,
9. infectious skin lesion at the site of the injection.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-11-13 (Actual); Primary Completion 2019-11-11 (Estimated); Study Completion 2019-11-13 (Estimated)

PRIMARY OUTCOMES:
Pain reduction after botox injection subjective | Change in clenching after 2,8,16,48 weeks
  Visual pain scale with a score from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Baraa abdulrahman, BDS, Principal Investigator — Riyadh Colleges of Dentistry and Pharmacy
Locations (1):
- Riyadh Elm University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No